CLINICAL TRIAL: NCT04831229
Title: The Influence of Interactive Media on Child Development in Children From 24 to 36 Months of Age: Protocol of a Randomized Controlled Clinical Trial
Brief Title: The Influence of Interactive Media on Child Development in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4.035.263; RBR-8j3tzw (Other: https://ensaiosclinicos.gov.br/rg/RBR-8j3tzw)
Record Dates: First submitted 2021-03-25; First posted 2021-04-05 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-01

CONDITIONS: Child Development
Keywords: Child Development; Tablet; Interactive Tutorial

STUDY DESIGN:
Intervention Model Description: We propose an RCT with 64 children aged 24 to 36 months and their parents. Measures of cognitive, motor and language development through the Bayley III Scale and Auditory Vocabulary Test. For follow-up purposes, parents will be asked to complete the Daily Record Board. Children will be randomly randomized into two groups: Active Interactive Media Group: children will use the media actively (games) and Passive Interactive Media Group: children will use the media passively (content viewing). Both groups will participate in the intervention for 30 minutes, three times a week, for 16 weeks. After this period, children will be reassessed for cognitive, language and fine motor development, receptive vocabulary and analysis of the Daily Record Board.
Who Masked: Participant
Masking Description: Randomization will be carried out by means of a simple drawing where an independent researcher, not involved in the intervention or evaluation of the participants, will allocate the participants and it will be hidden using opaque and closed envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Interactive Media Group (Active Comparator): AIMG children will perform active activities on the interactive tablet media. The games and applications that will be used during this intervention were selected through a search in the online application store compatible with the tablet used during the intervention (Google Play). The search term used was "games for children aged 2 to 3 years" and they were analyzed for the following criteria: (1) interactivity: critical thinking, active participation, decision making; (2) learning: activities that stimulate cognitive development, fine motor, receptive language, expressive and social-emotional language (see table 1 to view activities); (3) suitability: age, period of development, multiple domains and (4) results: challenging activity, not frustrating, providing feedback
  Interventions: Other: Children will perform activities on interactive tablet; Other: Children will perform passive on interactive tablet
- Passive Interactive Media Group (Active Comparator): PIMG children will go to the intervention room where they will use interactive tablet media in passive activities, such as: watching videos and children's stories that they often watch at home. This survey will be possible thanks to the questionnaire on the Use of Interactive Media where parents will list which drawings, stories and videos children use to watch.
  Interventions: Other: Children will perform activities on interactive tablet; Other: Children will perform passive on interactive tablet

INTERVENTIONS:
Other: Children will perform activities on interactive tablet — AIMG will actively perform activities with user interaction with the equipment through touch or verbal response. Both groups will have a total of 48 intervention sessions.
  Other Names: active interactive tablet
Other: Children will perform passive on interactive tablet — The PIMG is just a spectator, having contact with the equipment only when switching on / off, "play" / pause ". Both groups will have a total of 48 intervention sessions.
  Other Names: Passive interactive tablet

SUMMARY:
Introduction: In the last decade the prevalence of the use of interactive media (smartphone, tablet) by children has grown worldwide. However, it is not yet known what its effects are on the development of children in early childhood and whether the form of use (passive or active) influences this practice. In view of this, the present study aims to assess, through a randomized clinical trial (RCT), whether the form of use of mobile interactive media interferes with the Methods: The investigators propose an RCT with 64 children aged 24 to 36 months and their parents. Initially, identification, information about the child and history of media use will be carried out through the Questionnaire on the Use of Interactive Media, economic classification (Brazil Economic Classification Criterion). Then, the quality of the school environment (Infant / Toddler Environment Rating Scale) will be observed and, finally, measures of cognitive, motor and language development through the Bayley III Scale and Auditory Vocabulary Test. For follow-up purposes, parents will be asked to complete the Daily Record Board. Children will be randomly randomized into two groups: Active Interactive Media Group: children will use the media actively (games) and Passive Interactive Media Group: children will use the media passively (content viewing). Both groups will participate in the intervention for 30 minutes, three times a week, for 16 weeks. After this period, children will be reassessed for cognitive, language and fine motor development, receptive vocabulary and analysis of the Daily Record Board.

Discussion: The results can provide (1) information on which form of use has the most benefits for children (2) guide parents, educators and health professionals on how to offer interactive media.

Trial registration: This clinical trial was submitted to and approved by the Research Ethics Committee of Universidade Federal dos Vales do Jequitinhonha e Mucuri (CAAE 29490420.9.0000.5108). The complete protocol was registered in the Clinical Trials REBEC ( https://ensaiosclinicos.gov.br) under number RBR-8j3tzw Keywords: Child Development, Tablet, Interactive Tutorial, Clinical Trial.

DETAILED DESCRIPTION:
The interactive media has different modes and levels of interactivity, being considered the use of active mode, when the child uses it with a high level of interactivity, performing tasks such as dragging, rotating and zooming on an object (as in games) or mode passive, when participants have a low level of interactivity, participants only understand the display of screen content and basic activities such as touching specific objects (eg play / pause when viewing videos and stories). The growth in the use of interactive media is mainly attributed to greater ease of access, due to its portability, as they are light, mobile and intuitive, being used from moments of leisure and entertainment to educational learning.

Both groups will receive interventions with the Interactive Tablet Media for 30 minutes, three times a week for a period of 16 weeks. The interventions will be carried out in an environment provided by the educational institution.

In the week before the start of the interventions, specific training will be carried out (on / off, ringing, double-tapping, increasing / decreasing, holding, increasing / decreasing volume) on the use of the equipment with the participating children. Children who are not included or who are excluded will remain in their classrooms carrying out activities already provided for in the institutional calendar.

Physiotherapists and physiotherapy students will be in the rooms conducting the interventions and elucidating possible doubts that may arise regarding the handling of the equipment.

Experimental Intervention 1 AIMG children will perform active activities on the interactive tablet media. The games and applications that will be used during this intervention were selected through a search in the online application store compatible with the tablet used during the intervention (Google Play). The search term used was "games for children aged 2 to 3 years" and they were analyzed for the following criteria: (1) interactivity: critical thinking, active participation, decision making; (2) learning: activities that stimulate cognitive development, fine motor, receptive language, expressive and social-emotional language (see table 1 to view activities); (3) suitability: age, period of development, multiple domains and (4) results: challenging activity, not frustrating, providing feedback.

Experimental Intervention 2 PIMG children will go to the intervention room where they will use interactive tablet media in passive activities, such as: watching videos and children's stories that they often watch at home. This survey will be possible thanks to the questionnaire on the Use of Interactive Media where parents will list which drawings, stories and videos children use to watch.

Treatment Contrast The main difference between the types of interventions is the mode of use and the level of interactivity of the interactive media, where the AIMG actively performs activities, that is, there is user interaction with the equipment through touch or verbal response and the performance of activities like rotating an object, dragging and zooming. PIMG is not the same, the user is just a spectator, having contact with the equipment only when switching on / off, choosing the content, performing activities such as increasing / decreasing the volume and touching certain specific objects such as giving "play" / pause ". Both groups will have a total of 48 intervention sessions.

Sample Size Calculation The G.Power 3.1® statistical program was used to determine the number of children. The sample size was based on the study by Huber and collaborators (2018) with results from the comparison of executive function tests in Australian children aged 24 to 48 months. For the trial, 64 children and their parents or guardians will be needed (n = 64). Participants will be randomly randomized into two groups: active interactive media group (n = 32) and passive interactive media group (n = 32), considering an independent t test with 80% power (beta error, type I), equal alpha at 0.05 and effect size of 0.63.

Data Management Plan Personal, demographic and economic data will be collected only once, before interventions start. Each child will be identified by code using the initial CMEI of origin and ascending order of numbering. This identification will be carried out by a person who will not participate in any phase of the research and will be stored in a safe place.

The data generated after evaluation will be analyzed and displayed in graphs, tables or images. They will be saved and stored on the computers of the main researchers, password protected, and on online platforms and will be accessed through common software. Data that is available on paper will be kept in a key office. It is important to note that all data will be treated confidentially.

The data will be preserved for at least five years after the end of the research by the responsible physiotherapist (SG), who will be closely supervised by the supervising professor (JS). If the project is discontinued by the responsible physiotherapist, the supervising professor will assume the role of the person responsible for the project at the Federal University of Vallyes do Jequitinhonha and Mucuri, Campus JK. Responsibility and decision making will be signed between all members of the project team in a homogeneous manner, always ensuring the security and quality of the data.

Data analysis A specific database will be elaborated in the Software SPSS22.0 (Statistical Package for the Social Sciences) in which specific research data will be allocated. For purposes of descriptive analysis, the frequency distribution of the categorical variables involved in the study evaluation and analysis of measures of central tendency and dispersion of continuous variables will be carried out. The normality of the data will be tested using the Kolmogorov-Smirnov test. For statistical analysis, in the case of parametric distribution, paired T tests will be used to compare the scores of the Bayley Test intragroup in the pre and post intervention moments with media. The student T test will be used to compare between the AIMG and PIMG groups. In case of non-parametric distribution, the Mann-Whitney and Kruskal-Wallis tests will be used. The significance level of 5% will be considered. All children in the groups will be reassessed, as an intention-to-treat analysis will be performed. This strategy analyzes the data of all participants included in the group for which they were selected, regardless of whether they completed the intervention.

Shielding In all phases of the project, care with blinding will be taken and supervised. Initially, as previously mentioned, the randomization of the participants will be blinded because it will be carried out by a person without involvement in the research. Assessors will also be blinded as they will not have access to which group the child and their parents are participating in and the same is identical for the groups. In the case of participants and physiotherapists and physiotherapy students who are connected to the intervention, blinding will be carried out as far as possible. One of the measures to be taken to avoid contact and contamination between groups is to carry out the intervention at different times. Physiotherapists and physiotherapy students involved in the treatment of AIMG will not be involved in providing PIMG intervention and vice versa. Outcome evaluators (statisticians) will also be completely blinded.

Ethic This study will be carried out in accordance with the Declaration of Helsinki. It was submitted and approved by the Research Ethics Committee (REC) of the Federal University of the Valleys of Jequitinhonha and Mucuri (UFVJM). The complete protocol will be registered in the Clinical Trials and in the Brazilian Registry of Clinical Trials. Participants will be asked for consent prior to any project related procedures.

This work was carried out with the support of the Coordination for the Improvement of Higher Education Personnel - Brazil (CAPES) - Financing Code and by the Research Support Foundation of the State of Minas Gerais - FAPEMIG (CDS - APQ-01887-17). Funders will not influence any decision making about the conduct of the study and will have no relationship with the manuscripts from the study

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are considered: children aged 24 to 36 months regularly enrolled in the Municipal Children's Education Centers (CMEIS);
* Participating in the study, children with limited experiences in the use of interactive media, <420 minutes / week or 60 minutes / day, which is within the recommendations of the Brazilian Society of Pediatrics (2019) and participation in research authorized and consented by parents or guardians. Being able to handle a tablet.

Exclusion criteria include: hildren with neurological disorders such as cerebral palsy or syndromes that affect cognitive, linguistic and motor aspects, autism, moderate to severe hearing loss, mental or psychiatric disorders, prematurity and low birth weight.

* children with neurological disorders such as cerebral palsy or syndromes that affect cognitive, linguistic and motor aspects, autism, moderate to severe hearing loss, mental or psychiatric disorders, prematurity and low birth weight.

Ages: 24 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2021-08-21 (Estimated); Primary Completion 2022-08-21 (Estimated); Study Completion 2023-08-21 (Estimated)

PRIMARY OUTCOMES:
Cognitive development was chosen as a primary outcome measure, as interactive media it is known to be affected by interactive media. | Tests performed before the intervention
  To assess development in the cognitive domain, the Bayley III scale will be used, which assesses children from one to 42 months of age. The total score is converted into a balanced score and / or composed using tables provided in the manual. The composite score is based on age standards, where the child is rated from 40 to 160. The average score is 100, with ± 15 points standard deviation. This score will classify children into ranges: much higher (> 130 points), higher (between 129 to 120 points), above average (119 to 110 points), average (109 to 90 points), below average (89 at 80 points), borderline (79 to 70 points) and extremely low (69 or less points).
Motor development was chosen as a primary outcome measure, as interactive media it is known to be affected by interactive media. | Tests performed before the intervention
  To assess development in the Motor domain, the Bayley III scale will be used, which assesses children from one to 42 months of age. The total score is converted into a balanced score and / or composed using tables provided in the manual. The composite score is based on age standards, where the child is rated from 40 to 160. The average score is 100, with ± 15 points standard deviation. This score will classify children into ranges: much higher (> 130 points), higher (between 129 to 120 points), above average (119 to 110 points), average (109 to 90 points), below average (89 at 80 points), borderline (79 to 70 points) and extremely low (69 or less points).
Language development was chosen as a primary outcome measure. | Tests performed before the intervention
  The assess the receptive vocabulary of children, a validated instrument, the Auditory Vocabulary Test (TVAud - A33o), will also be used.According to age and score, children will be classified as follows: 2 year old children: medium level (17 and 28 points); low (12 and 16 points), very low (6 and 11 points) and high (29 and 33 points). 3-year-old children: medium level (24 and 31 points), low (21 and 23 points), very low (17 and 20 points) and high (31 and 33 points).
Change Cognitive development was chosen as a primary outcome measure, as interactive media it is known to be affected by interactive media. | Tests performed after 16 weeks of intervention
  To assess development in cognitive, motor and linguistic domains, the Bayley III scale will be used, which assesses children from one to 42 months of age in order to identify developmental delay. The score can be converted into balanced scores and / or composed through the use of tables provided in the manual. The approximate duration of the scale application is 50 minutes. The Bayley III test is the gold standard for development assessment and validated for the Brazilian population.
Change Motor development was chosen as a primary outcome measure, as interactive media it is known to be affected by interactive media. | Tests performed after 16 weeks of intervention
  To assess development in motor domains, the Bayley III scale will be used, which assesses children from one to 42 months of age in order to identify developmental delay. The score can be converted into balanced scores and / or composed through the use of tables provided in the manual. The approximate duration of the scale application is 50 minutes. The Bayley III test is the gold standard for development assessment and validated for the Brazilian population.
Change language development was chosen as a primary outcome measure. | Tests performed after 16 weeks of intervention
  o assess the receptive vocabulary of children, a validated instrument, the Auditory Vocabulary Test (TVAud - A33o), will also be used.

SECONDARY OUTCOMES:
For the purpose of identifying and controlling variables that may interfere with child development- For economic classification | Tests performed before the intervention
  For economic classification, the Brazilian Economic Classification Criterion (CCBB) of the Brazilian Association of Research Companies (ABEP) 2019, based on this score, the family's economic.
The quality of the school environment children experience | Tests performed before the intervention
  The quality of the school environment children experience, the Infant/Toddler Environment Rating Scale (ITERS-R) will be used. To assess opportunities children have at home, the Affordances in the Home Environment for Motor Development (AHEMD) will be used. The scale has 39 items distributed in seven subscales that are indicators of quality: (1) space and furniture; (2) personal care routine; (3) speaking and understanding; (4) activities; (5) interaction; (6) program structure; (7) parents and staff. In the environment to be evaluated in the early childhood education institution.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana D Nunes, Dr, Study Director — Federal University of the Valleys of Jequitinhonha and Mucuri

IPD SHARING:
Plan to Share IPD: Yes
Personal, demographic and economic data will be collected only once, before interventions start. Each child will be identified by code using the initial CMEI of origin and ascending order of numbering. This identification will be carried out by a person who will not participate in any phase of the research and will be stored in a safe place.
  The data generated after evaluation will be analyzed and displayed in graphs, tables or images. They will be saved and stored on the computers of the main researchers, password protected, and on online platforms and will be accessed through common software. Data that is available on paper will be kept in a key office. It is important to note that all data will be treated confidentially.
  The data will be preserved for at least five years after the end of the research by the responsible physiotherapist (SG), who will be closely supervised by the supervising professor (JS)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years
Access Criteria: Request to the responsible physiotherapist

REFERENCES:
- [Background] Radesky JS, Christakis DA. Increased Screen Time: Implications for Early Childhood Development and Behavior. Pediatr Clin North Am. 2016 Oct;63(5):827-39. doi: 10.1016/j.pcl.2016.06.006. PMID 27565361
- [Background] Bernard JY, Padmapriya N, Chen B, Cai S, Tan KH, Yap F, Shek L, Chong YS, Gluckman PD, Godfrey KM, Kramer MS, Saw SM, Muller-Riemenschneider F. Predictors of screen viewing time in young Singaporean children: the GUSTO cohort. Int J Behav Nutr Phys Act. 2017 Sep 5;14(1):112. doi: 10.1186/s12966-017-0562-3. PMID 28870219
- [Background] 3. Common Sense Media. The common sense census: media use by kids age zero to eight. 2017.
- [Background] 4. Piñeiro ES, González CR. Repercusión de la interactividad y los nuevos medios de comunicación en los procesos educativos. Investigación y Postgrado. 2006;21(1):187-209.
- [Background] 5. Agnaldo Pedra A, Mayer RE Albertin AL. Role of Interactivity in Learning from Engineering Animations. Appl. Cognit. Psychol.2015. p. 614-20.
- [Background] 6. Rideout V. Learning at home: families' educational media use in America. The Joan Ganz Cooney Center: New York; 2014.
- [Background] 7. Merchant G. Keep taking the tablets : iPads, story apps and early literacy. Australian Journal of Language and Literacy. 2015;38:3-11.
- [Background] 8. Piotrowski JT, Krcmar M. Reading with hotspots: Young children's responses to touchscreenstories. Computers in Human Behavior [Internet]. 2017; 70(0747-5632):[328-34 pp.].
- [Background] Wu CS, Fowler C, Lam WY, Wong HT, Wong CH, Yuen Loke A. Parenting approaches and digital technology use of preschool age children in a Chinese community. Ital J Pediatr. 2014 May 7;40:44. doi: 10.1186/1824-7288-40-44. PMID 24887105
- [Background] COUNCIL ON COMMUNICATIONS AND MEDIA. Media and Young Minds. Pediatrics. 2016 Nov;138(5):e20162591. doi: 10.1542/peds.2016-2591. PMID 27940793
- [Background] Wood E, Petkovski M, De Pasquale D, Gottardo A, Evans MA, Savage RS. Parent Scaffolding of Young Children When Engaged with Mobile Technology. Front Psychol. 2016 May 10;7:690. doi: 10.3389/fpsyg.2016.00690. eCollection 2016. PMID 27242603
- [Background] Guedes SDC, Morais RLS, Santos LR, Leite HR, Nobre JNP, Santos JN. CHILDREN'S USE OF INTERACTIVE MEDIA IN EARLY CHILDHOOD - AN EPIDEMIOLOGICAL STUDY. Rev Paul Pediatr. 2019 Nov 25;38:e2018165. doi: 10.1590/1984-0462/2020/38/2018165. eCollection 2020. PMID 31778410
- [Background] 14. Ré AHN. Crescimento, maturação e desenvolvimento na infância e adolescência: Implicações para o esporte. Motricidade [Internet]. 2011; 7:55-67. Available from: http://www.scielo.mec.pt/pdf/mot/v7n3/v7n3a08.pdf.
- [Background] Daelmans B, Darmstadt GL, Lombardi J, Black MM, Britto PR, Lye S, Dua T, Bhutta ZA, Richter LM; Lancet Early Childhood Development Series Steering Committee. Early childhood development: the foundation of sustainable development. Lancet. 2017 Jan 7;389(10064):9-11. doi: 10.1016/S0140-6736(16)31659-2. Epub 2016 Oct 4. No abstract available. PMID 27717607
- [Background] 16. Pediatria SBd. Saúde da Criança e Adolescentes na Era Digital. Manual de Orientação. In: Adolescência Dd, editor. 2016.
- [Background] 17. Calder N. Apps: Appropriate, Applicable, and Appealing? 2014. In: Digital Games and Mathematics Learning: Potential, Promises and Pitfalls [Internet]. Springer; 233-50.
- [Background] 18. Huber B, Tarasuik J, Antoniou MN, Garrett C, Bowe SJ, Swinburne JK, et al. Young children's transfer of learning from a touchscreen device. Comput Human Behav [Internet]. 2016; 56: 56-64. Available from: https://www.sciencedirect.com/science/article/pii/S0747563215302259.
- [Background] 19. Hallstedt H, Ghaderi TKA. Short and Long-Term Effects of a Mathematics Tablet Intervention for Low Performing Second Graders. Journal of Educational Psychology [Internet]. 2018; 110:1127-48.
- [Background] Huber B, Yeates M, Meyer D, Fleckhammer L, Kaufman J. The effects of screen media content on young children's executive functioning. J Exp Child Psychol. 2018 Jun;170:72-85. doi: 10.1016/j.jecp.2018.01.006. Epub 2018 Feb 12. PMID 29448235
- [Background] 21. Papadakis S, Kalogiannakis M, Zaranis, N. The effectiveness of computer and tablet assisted intervention in early childhood students' understanding of numbers. An empirical study conducted in Greece. Educ Inf Technol [Internet]. 2018; 23:1849-71.
- [Background] 22. LinC-C. Learning English with electronic textbooks on tablet PCs. Interactive Learning Environments [Internet]. 2016; (1744-5191).
- [Background] 23. Ebrahimzadeh M. Readers, Players, and Watchers: EFL Students' Vocabulary Acquisition through Digital Video Games. Canadian Center of Science and Education [Internet]. 2017; 10, 1-18.
- [Background] Dempsey AG, Barton AK, Duncan AF. Differences in Performance on Developmental Tasks in Young Children Across Digital and Paper-Based Modalities: A Feasibility Trial. J Dev Behav Pediatr. 2018 Dec;39(9):726-735. doi: 10.1097/DBP.0000000000000618. PMID 30418301
- [Background] Klop D, Marais L, Msindwana A, De Wet F. Learning new words from an interactive electronic storybook intervention. S Afr J Commun Disord. 2018 Sep 13;65(1):e1-e8. doi: 10.4102/sajcd.v65i1.601. PMID 30326711
- [Background] 26. Labrensz J, Ayebo A. Effects of Personal Learning Devices and Their Usageson Student Learning and Engagement. Jl of Computers in Mathematics and Science Teaching [Internet]. 2018; 37:193-216.
- [Background] Barnett LM, Ridgers ND, Reynolds J, Hanna L, Salmon J. Playing Active Video Games may not develop movement skills: An intervention trial. Prev Med Rep. 2015 Aug 13;2:673-8. doi: 10.1016/j.pmedr.2015.08.007. eCollection 2015. PMID 26844136
- [Background] Johnson TM, Ridgers ND, Hulteen RM, Mellecker RR, Barnett LM. Does playing a sports active video game improve young children's ball skill competence? J Sci Med Sport. 2016 May;19(5):432-6. doi: 10.1016/j.jsams.2015.05.002. Epub 2015 May 15. PMID 26050626
- [Background] 29. Vernadakis N, Papastergiou M, Zetou E, Antoniou P. The impact of an exergame-based intervention on children's fundamental motor skills. Computers & Education [Internet]. 2015; 83:90-102.
- [Background] Souto PHS, Santos JN, Leite HR, Hadders-Algra M, Guedes SC, Nobre JNP, Santos LR, Morais RLS. Tablet Use in Young Children is Associated with Advanced Fine Motor Skills. J Mot Behav. 2020;52(2):196-203. doi: 10.1080/00222895.2019.1602505. Epub 2019 Apr 22. PMID 31007146
- [Background] 31. Neumann MM. Using tablets and apps to enhance emergent literacy skills in young children. Early Childhood Research Quarterly [Internet]. 2018; 42:239-46.
- [Background] 32. Nortcliffe A, Middleton A. The innovative use of personal smart devices by students to support their learning. . In: Wankel L, Blessinger P, editors. Increasing student engagement and retention using mobile applications: Smartphones, Skype and texting technologies Emerald: Cutting Edge Technologies in Higher Education; 2013. p. 175-208.
- [Background] Poitras VJ, Gray CE, Janssen X, Aubert S, Carson V, Faulkner G, Goldfield GS, Reilly JJ, Sampson M, Tremblay MS. Systematic review of the relationships between sedentary behaviour and health indicators in the early years (0-4 years). BMC Public Health. 2017 Nov 20;17(Suppl 5):868. doi: 10.1186/s12889-017-4849-8. PMID 29219092
- [Background] 34. Bayley N. Bayley scales of infant and and toddller development: technical manual. 3, editor. San Antonio: Pearson; 2006.
- [Background] 35. Madaschi V, Mecca TP, Macedo EC, Paula CS. Escalas Bayley-III de Desenvolvimento Infantil: Adaptação Transcultural e Propriedades Psicométricas. Paidéia (Ribeirão Preto) [online]. 2016;26(64):189-97.
- [Background] Johnson S, Marlow N. Developmental screen or developmental testing? Early Hum Dev. 2006 Mar;82(3):173-83. doi: 10.1016/j.earlhumdev.2006.01.008. Epub 2006 Feb 28. PMID 16504424
- [Background] 37. Capovilla FC, Negrão VB, Damazio M. Teste de Vocabulário Auditivo e Teste de Vocabulário Expressivo. . São Paulo, SP: Memnon Edições Científicas Ltda 2011.
- [Background] 38. ABEP. Brazilian Economic Classification Criterion. 2018.
- [Background] 39. Carvalho AM. Qualidade em Ambientes de um Programa de Educação Infantil. . Psicologia: Teoria e Pesquisa [Internet]. 2008; 24:269-77.
- [Background] 40. Kaarby KME, Tandberg C. ITERS-R as a tool for improving quality in Norwegian ECEC settings: A critical reflection. . Journal of the European Teacher Education Network [Internet]. 2018; 13: 58-70.
- [Background] 41. Gennaro LRM, Gil MSCA. Análise teórica de itens de uma escala Americana para avaliação do atendimento em creches inclusivas brasileiras. Educação Especial; 2012. p. 531-44.
- [Background] 42. Amaro LLdM, Pinto SA, Morais RLdS, Tolentino JA, Felício LR, Camargos ACR, et al. Desenvolvimento infantil: comparação entre crianças que frequentam ou não creches públicas . . Journal of Human Growth and Development; 2015.
- [Background] 43. Rodrigues L, Gabbard C. Avaliação das oportunidades de estimulação motora presentes na casa familiar: projecto affordances in the home environment for motor development. FMH ed. Lisboa: Desenvolvimento Motor da Criança.; 2007. p. 51-60.
- [Background] 44. U.S. Department of Health & Human Services. Interactive Head Start Early Learning Outcomes Framework: Ages Birth to Five [Available from: https://eclkc.ohs.acf.hhs.gov/interactive-head-start-early-learning-outcomes-framework-ages-birth-five
- See also: The complete protocol was registered in the Brazilian Registry of Clinical Trials -REBEC — https://ensaiosclinicos.gov.br/rg/RBR-8j3tzw
- Available data/document: Study Protocol: Registration platform REBEC — https://ensaiosclinicos.gov.br/rg/RBR-8j3tzw — Project registered at REBEC